CLINICAL TRIAL: NCT04589962
Title: SUrgical Versus PERcutaneous AXillary Artery International Registry A Physician-initiated, International, Multicentric, Retrospective, Observational, Voluntary Registry - SUPER AXA International Registry
Brief Title: SUrgical Versus PERcutaneous AXillary Artery International Registry
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Principal Investigator, IRCCS San Raffaele
Other Study IDs: SUPER AXAInternationalRegistry
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Surgical and the Percutaneous Approach to the Upper Extremity Access

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Percutaneous Group
  Interventions: Other: access axillary or brachial artery
- Surgical Group
  Interventions: Other: access axillary or brachial artery

INTERVENTIONS:
Other: access axillary or brachial artery — access to the axillary or brachial artery during Transcatheter Aortic Valve Implantation (TAVI), Fenestrated/Branched-Endovascular Aortic Repair (F/BEVAR), chimney-EVAR (Ch-EVAR) or visceral side branches stenting

SUMMARY:
The purpose of the Study is to compare the outcomes of the surgical and the percutaneous approach to the upper extremity access (axillary or brachial artery) during endovascular procedures on the aortic valve, the aorta, and its side branches.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a surgical or percutaneous access to the axillary or brachial artery during Transcatheter Aortic Valve Implantation (TAVI), Fenestrated/Branched-Endovascular Aortic Repair (F/BEVAR), chimney-EVAR (Ch-EVAR) or visceral side branches stenting, between January 2010 and May 2020
* Adult patients ≥18 years

Exclusion Criteria:

* Introducer sheath internal diameter (ID) used < 5F or > 22F
* Patient with previous surgical axillary access on the puncture side (Pacemaker excluded)
* Patient with subclavian / axillary / brachial occlusive disease with stenosis greater than 50%
* Patient with previous bypass surgery or stent placement in the vicinity of access site (ie. Axillary extracorporeal cannulation with, axillo-femoral bypass, patch (venous or synthetic repair of previous axillary access, etc)
* Bleeding diathesis or coagulopathy
* Patients with active systemic or cutaneous infection or inflammation
* Patients who are pregnant or lactating
* Patient younger than 18 years of age
* Patients who are morbidity obese (BMI > 40 Kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated between January 2010 and May 2020 for a condition involving the aortic valve or the aorta and/or its side branches with procedures requiring an upper extremity access at the level of the axillary or brachial artery
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
optimal hemostasis | 30 days
  Closure success rate of the procedure without any adjunctive procedures
vascular complications | 30 days
  freedom from major access vascular complications requiring adjunctive endovascular or open procedures
Incidence of permanent peripheral nerve injury | 30 days
  freedom from permanent peripheral nerve injury with functional compromise
stroke Incidence | periprocedural
  freedom from periprocedural stroke
Durability of vessel closure | 30 days
  freedom from secondary intervention at access site

CONTACTS AND LOCATIONS:
Overall Officials: Luca Bertoglio, MD, Principal Investigator — IRCCS San Raffaele Hospital
Locations (18):
- Ascension St John Hospital and Medical Center, Detroit, Michigan, United States
- Medical University of Vienna, Vienna, Austria
- Imelda Hospital, Bonheiden, Belgium
- Service de Chirurgie Thoracique et Cardiovasculaire, Rennes, France
- Germany (5):
  - University Hospital of Cologne, Cologne
  - Asklepios Klinik St. Georg, Hamburg
  - University Heart and Vascular Center Hamburg, Hamburg
  - University Hospital Hamburg-Eppendorf, Hamburg
  - University hospital Leipzig, Leipzig
- Italy (4):
  - IRCCS San Raffaele Hospital, Milan
  - IRCCS San Raffaele, Milan
  - S. Maria della Misericordia Hospital, Perugia
  - San Filippo Neri Hospital, Roma
- Spain (2):
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Álvaro Cunqueiro, Vigo
- Skåne University Hospital, Malmo, Sweden
- UniversitätsSpital Zürich, Zurich, Switzerland
- Nuffield Dept. of Clinical Neurosciences, University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mirza AK, Oderich GS, Sandri GA, Tenorio ER, Davila VJ, Karkkainen JM, Hofer J, Cha S. Outcomes of upper extremity access during fenestrated-branched endovascular aortic repair. J Vasc Surg. 2019 Mar;69(3):635-643. doi: 10.1016/j.jvs.2018.05.214. Epub 2018 Oct 24. PMID 30714569
- [Background] Branzan D, Steiner S, Haensig M, Scheinert D, Schmidt A. Percutaneous Axillary Artery Access for Endovascular Treatment of Complex Thoraco-abdominal Aortic Aneurysms. Eur J Vasc Endovasc Surg. 2019 Sep;58(3):344-349. doi: 10.1016/j.ejvs.2019.01.011. Epub 2019 Jul 30. PMID 31375342
- [Background] Malgor RD, Marques de Marino P, Verhoeven E, Katsargyris A. A systematic review of outcomes of upper extremity access for fenestrated and branched endovascular aortic repair. J Vasc Surg. 2020 May;71(5):1763-1770.e2. doi: 10.1016/j.jvs.2019.09.028. Epub 2019 Nov 15. PMID 31740188
- [Background] Deuschl F, Schofer N, Seiffert M, Hakmi S, Mizote I, Schaefer A, Schirmer J, Reichenspurner H, Blankenberg S, Conradi L, Schafer U. Direct percutaneous transaxillary implantation of a novel self-expandable transcatheter heart valve for aortic stenosis. Catheter Cardiovasc Interv. 2017 Dec 1;90(7):1167-1174. doi: 10.1002/ccd.26986. Epub 2017 Mar 15. PMID 28296065
- [Background] Schafer U, Deuschl F, Schofer N, Frerker C, Schmidt T, Kuck KH, Kreidel F, Schirmer J, Mizote I, Reichenspurner H, Blankenberg S, Treede H, Conradi L. Safety and efficacy of the percutaneous transaxillary access for transcatheter aortic valve implantation using various transcatheter heart valves in 100 consecutive patients. Int J Cardiol. 2017 Apr 1;232:247-254. doi: 10.1016/j.ijcard.2017.01.010. Epub 2017 Jan 7. PMID 28118931
- [Background] Frohlich GM, Baxter PD, Malkin CJ, Scott DJ, Moat NE, Hildick-Smith D, Cunningham D, MacCarthy PA, Trivedi U, de Belder MA, Ludman PF, Blackman DJ; National Institute for Cardiovascular Outcomes Research. Comparative survival after transapical, direct aortic, and subclavian transcatheter aortic valve implantation (data from the UK TAVI registry). Am J Cardiol. 2015 Nov 15;116(10):1555-9. doi: 10.1016/j.amjcard.2015.08.035. Epub 2015 Sep 3. PMID 26409640
- [Background] Arnett DM, Lee JC, Harms MA, Kearney KE, Ramos M, Smith BM, Anderson EC, Tayal R, McCabe JM. Caliber and fitness of the axillary artery as a conduit for large-bore cardiovascular procedures. Catheter Cardiovasc Interv. 2018 Jan 1;91(1):150-156. doi: 10.1002/ccd.27416. Epub 2017 Nov 11. PMID 29130612
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium (VARC)-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document (VARC-2). Eur J Cardiothorac Surg. 2012 Nov;42(5):S45-60. doi: 10.1093/ejcts/ezs533. Epub 2012 Oct 1. PMID 23026738
- [Background] Bertoglio L, Grandi A, Melloni A, Kahlberg A, Melissano G, Chiesa R. Percutaneous AXillary Artery (PAXA) Access at the First Segment During Fenestrated and Branched Endovascular Aortic Procedures. Eur J Vasc Endovasc Surg. 2020 Jun;59(6):929-938. doi: 10.1016/j.ejvs.2020.01.027. Epub 2020 Feb 20. PMID 32089506
- [Background] Schaefer A, Schirmer J, Schofer N, Schneeberger Y, Deuschl F, Blankenberg S, Reichenspurner H, Conradi L, Schafer U. Transaxillary transcatheter aortic valve implantation utilizing a novel vascular closure device with resorbable collagen material: a feasibility study. Clin Res Cardiol. 2019 Jul;108(7):779-786. doi: 10.1007/s00392-018-1407-z. Epub 2018 Dec 17. PMID 30560381
- [Background] De Palma R, Ruck A, Settergren M, Saleh N. Percutaneous axillary arteriotomy closure during transcatheter aortic valve replacement using the MANTA device. Catheter Cardiovasc Interv. 2018 Nov 1;92(5):998-1001. doi: 10.1002/ccd.27383. Epub 2017 Oct 25. PMID 29068128
- [Result] Puippe GD, Kobe A, Rancic Z, Pfiffner R, Lachat M, Pfammatter T. Safety of percutaneous axillary artery access with a suture-mediated closing device for parallel endograft aortic procedures - a retrospective pilot study. Vasa. 2018 Jun;47(4):311-317. doi: 10.1024/0301-1526/a000702. Epub 2018 Mar 27. PMID 29583101